CLINICAL TRIAL: NCT06464198
Title: Prospective Registry Study on the Implementation of Simultaneous Postoperative Radiochemotherapy for Salivary Gland Carcinomas of the Head and Neck Region
Status: Recruiting | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: GlandulaSimultan
Record Dates: First submitted 2024-06-12; First posted 2024-06-18 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-06

CONDITIONS: Locally Advanced Salivary Gland Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patient: Patients with locally advanced high-grade salivary gland carcinoma after oncological resection
  Interventions: Procedure: simultaneous postoperative radiochemotherapy

INTERVENTIONS:
Procedure: simultaneous postoperative radiochemotherapy — The efficacy and tolerability of simultaneous postoperative radiochemotherapy is being investigated.

SUMMARY:
This is a prospective registry study based on a standard therapy concept for postoperative simultaneous radiochemotherapy established in Erlangen and elsewhere. The efficacy and tolerability of simultaneous postoperative radiochemotherapy is being investigated. Patients with locally advanced high-grade salivary gland carcinoma after oncological resection are admitted.

ELIGIBILITY:
Inclusion Criteria:

* Salivary gland carcinomas of the major and minor salivary glands of the head and neck region
* High-grade histology
* Successful oncological resection with curative intent
* pT3-4 or pN1-3 or Pn1(perineural sheath infiltration) or pT1-2 with scarce or positive resection margin
* cM0
* Indication for postoperative combined radiochemotherapy (guideline-compliant radiochemotherapy; percutaneous radiotherapy up to a total dose of 64-72 Gy (depending on resection status), common chemotherapy regimens: Paclitaxel 135mg/m² KOF d1 and cisplatin 33mg/m² KOF d1-3, q d22 or paclitaxel 135mg/m² KOF d1, carboplatin AUC 1.5 KOF d1-3 or paclitaxel 50mg/m² KOF, carboplatin AUC2 d1,8,15, q d22 or paclitaxel 50mg/m²KOF and cisplatin 30mg/m² KOF d1,8,15, q d22, 4 cycles each).
* Patient age ≥18 years
* WHO performance score ≤ 1
* Signed patient information/consent form

Exclusion Criteria:

* Distant metastases
* Other cancer in the last 5 years prior to study inclusion (with the exception of: adequately treated skin cancer (except melanoma) or lentigo maligno or adequately treated carcinoma in situ, in each case without evidence of active disease).
* Previous chemotherapy or radiotherapy for salivary gland carcinoma
* Previous radiotherapy in the head and neck area
* Pre-existing uncontrolled disease that constitutes a contraindication to simultaneous combination chemotherapy (e.g. signs of acute heart failure, myocardial infarction within the last 6 months before the start of therapy, congestive heart failure, heart disease with New York Heart Association (NYHA) III or IV classification, active and therapy-resistant infection, pre-existing or concomitant immunodeficiency syndrome)
* Pregnancy and breastfeeding
* Fertile patients who cannot ensure effective contraception during and up to six months after combination therapy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced high-grade salivary gland carcinoma after oncological resection who fulfil the inclusion and exclusion criteria are included. Patients must be adequately informed about their diagnosis and about the nature, significance and scope of the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2036-06 (Estimated); Study Completion 2037-06 (Estimated)

PRIMARY OUTCOMES:
Creation of a database | 63 months (12 weeks therapy plus 5 years follow-up)
  Creation of a database of a representative homogeneously treated patient cohort with locally advanced salivary gland tumours receiving postoperative radiochemotherapy.

SECONDARY OUTCOMES:
Observation of Overall survival | 63 months (12 weeks therapy plus 5 years follow-up)
Observation of Disease-free survival | 63 months (12 weeks therapy plus 5 years follow-up)
Observation of Disease-specific survival | 63 months (12 weeks therapy plus 5 years follow-up)
Observation of Local recurrence-free survival | 63 months (12 weeks therapy plus 5 years follow-up)
Observation of Survival free of distant metastases | 63 months (12 weeks therapy plus 5 years follow-up)
Determination of toxicity | 63 months (12 weeks therapy plus 5 years follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Marlen Haderlein, PD Dr., Principal Investigator — Universitätsklinikum Erlangen, Strahlenklinik
Locations (1):
- Erlangen, Universitätsklinikum Strahlenklinik, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: No